CLINICAL TRIAL: NCT06865495
Title: Evaluating the Individual and Combined Effects of Hand Hygiene Promotion and Hardware Provision on Handwashing With Soap Behaviour in Urban and Peri-urban Lusaka, Zambia: a Factorial Randomised-controlled Trial
Brief Title: Evaluating the Individual and Combined Effects of Hand Hygiene Promotion and Hardware Provision on Handwashing With Soap in Lusaka, Zambia
Acronym: BCLab
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Centre for Infectious Disease Research in Zambia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 31387
Record Dates: First submitted 2025-02-24; First posted 2025-03-07 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-02

CONDITIONS: Handwashing Behaviour
Keywords: handwashing; hygiene; urban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Handwashing Hardware and Supply Provision (Experimental): Households in this arm will receive a locally available handwashing facility called the Kalingalinga bucket and be given supplies to make soapy water. They will receive a 3-month visit to check the facility is functioning.
  Interventions: Other: Handwashing Hardware and Supply Provision
- Hand Hygiene Behavioural Promotion (Experimental): Households in this arm will receive five bi-weekly educational visits, with a sixth follow-up visit four weeks later (6 visits in total).
  Interventions: Behavioral: Hand Hygiene Behavioural Promotion
- Handwashing Hardware and Supply Provision + Hand Hygiene Behavioural Promotion (Experimental): Households in this arm will receive both the hardware and supply provision and hand hygiene behavioural promotion interventions.
  Interventions: Other: Handwashing Hardware and Supply Provision; Behavioral: Hand Hygiene Behavioural Promotion
- Control (No Intervention): Households in this arm will receive no intervention during the study period. They will receive the most effective intervention combination after the study is complete.

INTERVENTIONS:
Other: Handwashing Hardware and Supply Provision — Households will be given a locally available handwashing facility called the Kalingalinga bucket. Intervention delivery workers will set-up the handwashing facility, and demonstrate how it works, including where to place soap on the stand. Households will also be given supplies and materials to make their own liquid soap from locally available soap products (soapy water). Discussions will also be held on HWF maintenance. This component of the intervention should take no longer than 30 minutes. Intervention delivery workers will return to households after three months (one visit) to ensure there are no issues with the handwashing station (e.g., broken stand or tap), to bring more liquid soap and to remind households how to make soapy water.
  Arms: Handwashing Hardware and Supply Provision; Handwashing Hardware and Supply Provision + Hand Hygiene Behavioural Promotion
Behavioral: Hand Hygiene Behavioural Promotion — The hand hygiene behavioural promotion intervention employs interactive storytelling and visual aids to promote handwashing with soap. Intervention delivery workers will act as storytellers, narrating stories about three characters with different handwashing habits.
  The intervention progresses through five bi-weekly visits, with a final sixth visit 4 weeks after the fifth visit. The 30-minute visits progress through different stages: (1) identifying behaviours, (2) understanding disease risks, (3) encouraging practical solutions and (4) promoting practice. The penultimate stage of the intervention focuses on reflection and commitment, encouraging participants to assess their behaviours and pledge to adopt improved hygiene practices. The final visit allows participants to reflect on the whole intervention and covers information participants would like to revisit.
  Arms: Hand Hygiene Behavioural Promotion; Handwashing Hardware and Supply Provision + Hand Hygiene Behavioural Promotion

SUMMARY:
The goal of this study is to assess the individual and combined effects of hand hygiene behavioural promotion and handwashing hardware and supply provision on handwashing with soap behaviour at handwashing opportunities in households in peri-urban communities in Lusaka, Zambia.

Households will be randomly allocated to one of the four groups: AB) Hand hygiene behavioural promotion + handwashing hardware and supply provision, A) handwashing hardware and supply provision only, B) hand hygiene behavioural promotion only or C) No intervention.

Researchers will compare handwashing behaviour between the four groups to see which is most effective.

DETAILED DESCRIPTION:
The study is a superiority, multi-arm, parallel group randomised-controlled trial. A total of 1800 households within five wards in Lusaka will be enrolled. Eligible households include households with at least one child under the age of 5, with no fixed handwashing facility, and at least one adult (18+) who can consent to the study. Households must also be permanent residents of the communities (i.e., expect to remain in the community for the next 3-6 months).

Households will be randomly assigned to one of four arms (450 households per arm) (1:1:1:1): (AB) hand hygiene behavioural promotion + handwashing hardware and supply provision, (A) handwashing hardware and supply provision only, (B) hand hygiene behavioural promotion only, (C) control group (receive most effective intervention after the study ends).

For households receiving the hardware and supply intervention, a handwashing facility with supplies to make liquid soap (soapy water) will be provided and left with households for six months, with a visit at 3-months to check the handwashing facility is functioning and to provide more soap supplies. For households receiving the hand hygiene behavioural promotion intervention, 5 bi-weekly household visits (30 minutes) will be conducted, with a sixth follow-up visit four weeks later, for a total of 6 planned "touch points".

Handwashing with soap (HWWS) at handwashing opportunities (before cooking, before eating, before feeding a child, before breastfeeding, after toilet use, after handling child/adult faeces or cleaning a child's bottom, after contact with animals and after coughing/sneezing) will be measured using 3-hour structured observations of one household member per household, conducted at baseline and endline (6-months are intervention delivery begins).

ELIGIBILITY:
Eligibility is assessed at the household level.

Inclusion Criteria:

* At least one adult (aged 18 or older) who can consent to the study on behalf of all members of the household.
* At least one child under the age of 5.

Exclusion Criteria:

* Already own a similar handwashing facility (e.g., sink, handwashing station).
* Not permanent residents of the selected community and/or plans to leave the community within the next 3-6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Handwashing with soap (HWWS) at all handwashing opportunities | Measured at baseline and endline (6-months after intervention delivery begins)
  The probability of HWWS within three minutes of any handwashing opportunity (before cooking, before eating, before feeding a child, before breastfeeding, after toilet use, after handling child/adult faeces or cleaning a child's bottom, after contact with animals and after coughing/sneezing) in the correct sequence (e.g., before or after the relevant opportunity); measured through direct observation of individual behaviour over a a three-hour observation period.

SECONDARY OUTCOMES:
Handwashing with soap (HWWS) at each specific handwashing opportunity. | Measured at baseline and endline (6-months after intervention delivery begins)
  The probability of HWWS at each specific handwashing opportunity (before cooking, before eating, before feeding a child, before breastfeeding, after toilet use, after handling child/adult faeces or cleaning a child's bottom, after contact with animals and after coughing/sneezing); measured through direct observation of individual behaviour over a a three-hour observation period.
Hand-rinsing measured as a three-level outcome: no action, hand-rinsing or handwashing with soap at all handwashing opportunities. | Measured at baseline and endline (6-months after intervention delivery begins)
  The probability of either HWWS, hand rinsing with water only, or taking no action within three minutes of any handwashing opportunity (before cooking, before eating, before feeding a child, before breastfeeding, after toilet use, after handling child/adult faeces or cleaning a child's bottom, after contact with animals and after coughing/sneezing) in the correct sequence (e.g., before or after the relevant opportunity); measured through direct observation of individual behaviour over a a three-hour observation period.
Handwashing Facility Presence | Measured at baseline and endline (6-months after intervention delivery begins)
  The probability that a household has a fully functional handwashing facility with water and soap present.
Handwashing knowledge and reported practice. | Measured at baseline and endline (6-months after intervention delivery begins)
  Knowledge: Number of opportunities (before cooking, before eating, before feeding a child, before breastfeeding, after toilet use, after handling child/adult faeces or cleaning a child's bottom, after contact with animals and after coughing/sneezing) for handwashing with soap correctly specified in response to the question "When do you think it is important to wash hands with soap?".
  Reported practice: Number of opportunities (before cooking, before eating, before feeding a child, before breastfeeding, after toilet use, after handling child/adult faeces or cleaning a child's bottom, after contact with animals and after coughing/sneezing) for handwashing with soap reported in response to the question "When did you wash your hands with soap yesterday?"
  Both questions assessed through survey of open-ended questions with pre-coded responses and multiple rounds of probing.

OTHER OUTCOMES:
Diarrhoeal Illness | Measured at baseline and endline (6-months after intervention delivery begins)
  The risk of self-reported diarrhoea at least once in the past 7 days according to WHO definition of diarrhoea - 3 or more loose stools in 24hrs. Measured through survey with primary respondents. Results will be stratified by age group.
Respiratory Illness | Measured at baseline and endline (6-months after intervention delivery begins)
  The risk of self-reported respiratory illness at least once in the past 7 days according to WHO definition of respiratory illness - coughing or difficulty breathing. Measured through survey with primary respondents. Results will be stratified by age group.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dreibelbis, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Centre for Infectious Disease Research in Zambia (CIDRZ), Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
All data will be fully anonymised and posted on a public repository for third party use. To completely anonymise the data prior to uploading it onto an open data site any information that holds the potential to identify the respondents will be redacted.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available within 2 years of endline data collection.
Access Criteria: To be determined.